CLINICAL TRIAL: NCT05076318
Title: Dysregulated Urea-synthesis at Terminal Uremia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dysregulated urea-synthesis
Record Dates: First submitted 2021-08-26; First posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-01

CONDITIONS: Urea Cycle Disorder; Uremia
MeSH Terms: conditions — Urea Cycle Disorders, Inborn; Uremia | interventions — Amino Acids

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alanine-infusion (Experimental): Alanine infusion taking place over a 3 hour period while monitorering metabolic changes in blood samples before and after dialysis
  Interventions: Other: Aminoacid, alanine-infusion

INTERVENTIONS:
Other: Aminoacid, alanine-infusion — During 3 hours, patient will receive alanine-infusion, while amino-acid and urea will be monitored by blood samples.

SUMMARY:
This project will examine the dysregulation of the urea cycle in patients with terminal uremia using a validated method named "Functional Hepatic Nitrogen Clearance"

ELIGIBILITY:
Inclusion Criteria:

* Age > or equal to 18 years
* Chronic hemodialysis during 3 months
* Patients with functioning arteriovenous-fistula assigned to "Center-Hemodialysis" at "Nyresygdomme, AUH Skejby"

Exclusion Criteria:

* Active infection
* Conditions with vomiting or diarrhea
* Diabetes
* Active disease being treated with chemotherapy, radiationtherapy, biologic- or similar treatments. Disease under observation can be included.
* Liver disease
* Vessels on the upper extremities not suited for cannulation
* Prednisolone treatment during the last 8 weeks
* Pregnancy
* BMI > or equal to 30 or < or equal to 18
* Physically or mentally condition that does not allow the project to be completed
* Language-difficulties that does not allow the project to be completed

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Urea synthesis rate during alanine infusion | 4 hours. 1 hour of blood sample measuring of baseline urea-synthesis rate and 3 hours of urea-synthesis rate during alanine-infusion
  Change in the synthesis of urea during a 3 hour period of alanine-infusion in pre and post hemodialysis patients. We will use a validated method named functional hepatic nitrogen clearance (FHNC) to evaluate the synthesis of urea. FHNC is calculated using the linear relation between urea nitrogen synthesis rate and blood-amino acid which is measured every hour. An estimated group of 10 dialysis patients will be included and compared to a clinical healthy group. The healthy group has also received alanine infusion and blood samples of urea and amino-acids has likewise been measured for every hour of infusion.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Aarhus, Aarhus N, Denmark